CLINICAL TRIAL: NCT04372862
Title: Comparison Between Serratus Anterior Plane Block and Erector Spinae Plane Block to Control Postmastectomy Pain
Brief Title: Comparison Between Serratus Anterior Plane Block and Erector Spinae Plane Block for Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ASPB vs ESBP for mastectomy
Record Dates: First submitted 2020-05-01; First posted 2020-05-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Postoperative Pain
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: prospective comparative randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus anterior plane block (Active Comparator): Serratus anterior plane block was performed in the supine position placing the ipsilateral upper limb in abduction 90 degrees position. Aiming to find the serratus anterior muscle the investigator identified the fifth rib in the mid-axillary line by the linear probe in the sagittal plane. The latissimus dorsi muscle (superficial and posterior), teres major muscle (superior) and serratus muscles (deep and inferior) were detected using ultrasound. The investigator penetrated the serratus anterior muscle by a 25 GA, 90 mm spinal needle in-plane concerning the ultrasound probe from superoanterior to posteroinferior to inject deep to it.
  Interventions: Procedure: Plane block
- Erector spinae plane block (Active Comparator): Erector spinae plane block was performed at lateral decubitus with the operation site up, the vertebrae were counted from cephalad to caudal direction until reaching T5 spinous process as the first palpable spinous process is C7. The ultrasound probe was placed vertically 3 cm lateral to the T5 spinous process. Three muscles were identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. The needle was introduced from superior to inferior direction in-plane until the tip lay deep to erector spinae muscle.
  Interventions: Procedure: Plane block

INTERVENTIONS:
Procedure: Plane block — Two different plane blocks to control post-mastectomy pain
  Other Names: Block

SUMMARY:
In this study, we are comparing two different techniques of plane blocks to control postoperative mastectomy pain serratus anterior plane block and erector spinae plane block, both are done with ultrasonic guidance We are recording the first time of analgesia request postoperatively as a primary outcome

ELIGIBILITY:
Inclusion Criteria:

* Female patient age 20 to 65
* ASA I, II
* Scheduled for mastectomy

Exclusion Criteria:

* Allergy to local anaesthetics
* Infection at the site of performing the block
* Morbidly obese patient of body mass index more than 40 kg/m2

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients of breast cancer operated for mastectomy
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
First time analgesia request | Postoperative up to 24 hours
  The first time the patient ask for analgesia to control postoperative pain

SECONDARY OUTCOMES:
Total analgesic consumption | Postoperative up to 24 hours
  The total calculated analgesics that were administered to control post operative pain
visual analogue scale | Every two hours for 24 hours postoperative
  A subjective method to measure pain, where 0=no pain and 10 = worst comprehensible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No